CLINICAL TRIAL: NCT01981278
Title: A Single-Dose, Open-Label, Randomized, 2-Way Crossover Pivotal Study to Assess Bioequivalence of a New Tapentadol Extended-Release (TRF) 250-mg Tablet With Respect to a Tapentadol Extended-Release (PR2) 250-mg Tablet Under Fasted Conditions in Healthy Subjects
Brief Title: A Study to Assess Bioequivalence of a New Tapentadol Extended-Release 250-mg Tablet With Respect to a Tapentadol Extended-Release 250-mg Tablet in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100458; R331333-PAI-1061 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Healthy; Tapentadol; Bioequivalence; Fasted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Tapentadol ER 250-mg tamper-resistant formulation (TRF) tablet will be administered as a single oral dose under fasted condition.
  Interventions: Drug: Tapentadol ER 250-mg TRF tablet
- Treatment B (Experimental): Tapentadol ER 250-mg prolonged-release formulation 2 (PR2) tablet will be administered as a single oral dose under fasted condition.
  Interventions: Drug: Tapentadol ER 250-mg PR2 tablet

INTERVENTIONS:
Drug: Tapentadol ER 250-mg TRF tablet — Participants will receive single oral dose of tapentadol ER 250-mg TRF tablet on Day 1 of each treatment period.
  Arms: Treatment A
Drug: Tapentadol ER 250-mg PR2 tablet — Participants will receive single oral dose of tapentadol PR2 250-mg tablet on Day 1 of each treatment period.
  Arms: Treatment B

SUMMARY:
The purpose of this study is to evaluate bioequivalence (scientific basis on which drugs with the same active ingredient(s) are compared) of a new tapentadol extended-release (ER) 250-mg tamper-resistant formulation (TRF) tablet to the current tapentadol ER 250-mg prolonged-release formulation 2 (PR2) tablet in healthy participants under fasted conditions.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center, randomized (the study medication is assigned by chance), 2-way crossover (method used to switch participants from one treatment arm to another in a clinical study) study of a single dose of 250-mg tapentadol. All participants will receive in randomized order the TRF tablet and PR2 tablet, both as a single dose of 250 mg tapentadol. Approximately 64 participants will be enrolled in the study. The study consists of 3 phases: a screening phase (within 2 to 21 days before the first study drug administration on Day 1 of Period 1), an open-label treatment phase consisting of 2 single-dose treatment periods. Treatment administrations will be separated by a washout period of 7 to 14 days. All participants will be randomly assigned to 1 of 2 possible treatment sequences and receive both of the following treatments, 1 in each period: Treatment A: tapentadol ER 250-mg TRF tablet, administered as a single oral dose under fasted condition and Treatment B: tapentadol ER 250-mg PR2 tablet, administered as a single oral dose under fasted condition. Safety will be evaluated by the assessment of adverse events, vital signs, physical examination, 12-lead electrocardiogram, and clinical laboratory tests which will be monitored throughout the study. The duration of participation in the study for an individual participant will be up to 5.5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study, are willing to participate in the study, and are willing to adhere to the prohibitions and restrictions specified in the protocol
* Healthy on the basis of pre-study physical examination, medical history, 12-lead electrocardiogram, vital signs, and clinical laboratory parameters performed within 21 days before study drug administration
* Women must have a negative serum human chorionic gonadotropin (hCG) pregnancy test at screening and on Day -1 of each treatment period
* Must agree to use an adequate contraception method and to not donate sperm during the study and for 3 months after receiving the last dose of study medication
* Body mass index (BMI) (weight [kg]/height [m2]) between 20 and 28 kg/m2, inclusive, and body weight not less than 50 kg

Exclusion Criteria:

* History of seizure disorder or epilepsy or mild or moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm within 1 year of screening, or severe traumatic brain injury within 15 years of screening, or severe traumatic brain injury resulting in ongoing sequelae suggesting transient changes in consciousness or symptoms
* History of a gastrointestinal disease affecting absorption, gastric surgery or history of or current significant medical illness including cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders, lipid abnormalities, significant pulmonary disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection
* History of clinically significant allergies, especially known hypersensitivity/intolerance or contraindications to opioids, opioid antagonists (eg, naloxone), benzodiazepines (eg, diazepam, clonazepam, lorazepam), any study drug formulation component, any of the excipients of the formulation, or heparin
* Women who plan to become pregnant during the study, or who are breast-feeding
* Positive test for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C antibodies

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of tapentadol | Predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  Cmax is defined as maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Time at Last Observed Quantifiable Concentration (AUClast) of tapentadol | Predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  AUClast is area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of tapentadol | Predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of tapentadol | Predose, and 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 36, 48 hours post-dose
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 5.5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C.Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Lincoln, Nebraska, United States